CLINICAL TRIAL: NCT02484183
Title: Effectiveness of Bubble Continuous Positive Airway Pressure (CPAP) in Reducing Childhood Pneumonia Mortality in Malawi
Brief Title: CPAP Improving Mortality for Pneumonia in African Children Trial
Acronym: IMPACT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: By Data Safety and Monitoring Board after second interim analysis and follow-up safety check.
Sponsor: Johns Hopkins University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Ministry of Health and Population, Malawi (Other Government); Children's Hospital Medical Center, Cincinnati (Other); University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00055734
Record Dates: First submitted 2015-06-23; First posted 2015-06-29 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Pneumonia; Human Immunodeficiency Virus (HIV); Malnutrition; Hypoxemia
Keywords: bubble continuous positive airway pressure (CPAP); pneumonia; Human Immunodeficiency Virus (HIV); malnutrition; Malawi; Africa; Noninvasive Ventilation; child; pediatric; hypoxemia
MeSH Terms: conditions — Pneumonia; Acquired Immunodeficiency Syndrome; Malnutrition; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-flow oxygen (No Intervention): Low-flow oxygen supplementation if respiratory danger signs are present or if their oxygen saturation is <90%. Respiratory danger signs include any of the following: grunting, severe chest indrawing, very fast breathing (>70 breaths/minute if 1-11 months; >60 breaths/minute if 12-59 months), nasal flaring, stridor in a calm child, or apnea. Low-flow oxygen given by an oxygen concentrator with a nasal cannula. Low-flow is 0.5 liters per minute (LPM) for patients 1-2 months, and 1-2 LPM for patients 2-59 months. For 2-59 month olds oxygen can be increased to a maximum of 2 LPM to maintain a 90% saturation or treat respiratory danger signs.
- bubble CPAP (Experimental): Bubble continuous positive airway pressure (bCPAP) patients are eligible if respiratory danger signs are present or if oxygen saturation is <90%. bCPAP will be initiated at 7 centimeters (cm) water (H20) if 1-2 months of age or 8cm H20 if 2-59 months of age using the minimum oxygen flow necessary to achieve these pressures. Gradual weaning can be attempted after 24-48 hours of treatment. All changes will be followed by 60 minutes of monitoring.
  Interventions: Device: bubble continuous positive airway pressure (CPAP)

INTERVENTIONS:
Device: bubble continuous positive airway pressure (CPAP) — This study will use an Airsep® oxygen concentrator and a Fisher & Paykel Bubble CPAP (bCPAP) system to deliver bCPAP. The Airsep® machine is connected to the Fischer & Paykel Bubble CPAP system and the CPAP delivers pressure and oxygen to the patient with appropriately sized masks and tubing. The Fischer & Paykel Bubble CPAP system can deliver up to 10 centimeters (cm) water (H20) pressure. Since an oxygen concentrator is being used as the flow driver of this bubble CPAP system patients receiving CPAP will therefore also be receiving 6-8 liters per minute (LPM) of concentrated oxygen flow. Per manufacturer specifications the Airsep oxygen concentrator delivers 90-97% fractional inspired oxygen concentration at the 6-8 LPM flows required to generate 4-10 cm H20 pressure.
  Other Names: Fisher and Paykel
  Arms: bubble CPAP

SUMMARY:
Pneumonia mortality rates in African countries like Malawi are high and increased further in children -exposed or infected with human immunodeficiency virus (HIV) as well as those that are severely malnourished or severely hypoxemic. Treatment innovations are needed. Bubble continuous positive airway pressure (bCPAP) improves oxygenation and ventilation and is a simple, relatively inexpensive adaptation of conventional continuous positive airway pressure potentially suitable for low-resource settings. bCPAP has been demonstrated to improve outcomes in neonates less than 1 month of age. Recently, a limited number of hospitals are using bCPAP to escalate pneumonia care for older African children failing standard treatment with antibiotics and oxygen. Supportive evidence for this approach is observational only. Quality randomized studies comparing bCPAP versus a standard-of-care control group that includes low-flow oxygen therapy and using a primary endpoint of mortality are not available in low-resource settings including high prevalence HIV countries like Malawi. Demonstrating a mortality benefit with bCPAP is needed to support further investment and scale up of bCPAP in the care of older Malawian children 1-59 months of age with World Health Organization (WHO) severe pneumonia complicated by HIV and/or malnutrition or severe hypoxemia.

With the full support of the Malawi Ministry of Health and in collaboration with external experts from Lilongwe Medical Relief Trust and Cincinnati Children's Hospital Medical Center investigators plan to address this critical evidence gap by conducting a randomized controlled study determining bCPAP outcomes, compared to the currently recommended standard of care endorsed by the WHO and Malawi national pneumonia guidelines, in hospitalized Malawian children with WHO-defined severe pneumonia complicated by a co-morbidity ((1) HIV-infection, (2) HIV-exposure without infection, (3) severely malnourished) or WHO pneumonia with severe hypoxemia and without a co-morbidity. The investigators hypothesize that bCPAP will reduce the mortality of Malawian children with WHO-defined severe pneumonia.

DETAILED DESCRIPTION:
Despite laudable reductions in global childhood mortality rates, pneumonia remains the second most frequent killer of children less than five years old worldwide. Nearly one million children succumbed to pneumonia in 2013, with greater than half of these deaths in Africa. In Malawi, which has a high prevalence of malnutrition and Human Immunodeficiency Virus (HIV) infection, pneumonia is a major cause of pediatric mortality. In patients with World Health Organization (WHO)-defined severe pneumonia, malnutrition, HIV-infection, and hypoxemia are the primary drivers of poor outcomes. In a recent analysis of 2001-2012 child pneumonia outcomes in Malawi the overall case fatality rate decreased from 15% to 4% except in children with severe malnutrition. The pneumonia mortality rate in malnourished children remained elevated at 15% despite antibiotics and increased access to supportive interventions like low-flow supplemental oxygen. In Malawian children with HIV-infection, WHO very severe pneumonia and severe malnutrition were the strongest predictors of death. Severe hypoxemic pneumonia may be as common in children as HIV-affected or severely malnourished cases, and may also have higher mortality than non HIV-affected, non-severely malnourished cases without severe hypoxemia. Non-invasive ventilation, already routinely used in industrialised countries, may provide an advanced treatment solution for certain patient populations such as children with WHO severe pneumonia complicated by severe malnutrition and/or HIV-infection or -exposure or severe hypoxemia.

Bubble continuous positive airway pressure (bCPAP) is non-invasive and is widely used for preterm neonatal respiratory failure in industrialised countries. Along with a flow generator, bCPAP uses a water column to deliver continuous positive pressure to a spontaneously breathing child. bCPAP is relatively inexpensive and requires little technical expertise compared with mechanical ventilation, but there is limited experience of bCPAP in resource-poor settings. Recently, small studies have explored its use in preterm neonates in Malawi. However, few studies have described its use in older infants and children, none of which included mortality as a primary endpoint and specially focused on the main drivers of poor pediatric pneumonia outcomes in southern Africa, HIV, malnutrition, and hypoxemia.

The investigators data using bCPAP in Malawian children with severe pneumonia suggest feasibility for implementation. The investigators have previously reported that using a bCPAP system derived from locally available, relatively inexpensive supplies has shown promise in the management of hospitalized HIV-infected children with pneumonia in Malawi. The investigators observational case series further delineates the outcomes of 77 Malawian children hospitalized at a tertiary referral facility with severe pneumonia who were treated with bCPAP. Nearly half were infants either infected or exposed to HIV or were severely malnourished. Although the mortality of this series of patients was 50.0%, bCPAP was initiated in this cohort only when patients were found to be failing standard treatment. The investigators estimated that more than 75% of these children would have been eligible for mechanical ventilation. In this proposed study the investigators will be initiating bCPAP earlier in the hospitalization prior to treatment failure. Unlike previous studies conducted at referral hospitals, the investigators will perform this study at the district hospital level where 80% of hospitalized child pneumonia cases are cared for in Malawi.

Although bCPAP is relatively inexpensive, scale-up in countries like Malawi with significant pneumonia burden and high HIV prevalence will require substantial resources to meet expected needs. In order to appropriately allocate precious resources and provide practical clinical guidance for healthcare providers who may use bCPAP, it is paramount to fully understand the utility of bCPAP treatment in this setting. To the investigators knowledge no bCPAP data using a control group with mortality as the primary outcome has been reporting in a similar generalized HIV epidemic African patient population 1-59 months of age. Data generated from this research will be additionally critical for formulating future studies that may include bCPAP refinements or exploration of other feasible modalities like high-flow nasal cannula or bi-level positive airway pressure. Therefore, the more rigorous methodology proposed here is warranted and supported by the Malawi Ministry of Health. If bCPAP proves an effective treatment modality for children hospitalized with WHO severe pneumonia, it is a simple technology that could be operationalized to help thousands of children with life-threatening pneumonia.

The investigators propose to address this critical evidence gap by conducting a randomized controlled study determining bCPAP outcomes, compared to the currently recommended standard of care endorsed by the WHO and Malawi Ministry of Health, in hospitalized Malawian children with WHO-defined severe pneumonia complicated by malnutrition and/or HIV-infection or -exposure, or severe hypoxemia.

RATIONALE

Quality randomized studies comparing bCPAP versus a standard-of-care control group that includes low-flow oxygen therapy and using a primary endpoint of mortality are not available in low-resource settings including high prevalence HIV countries like Malawi for children 1-59 months of age with severe pneumonia. Demonstrating a mortality benefit with bCPAP is needed to support further investment and scale up of bCPAP in the care of older Malawian children 1-59 months of age with World Health Organization (WHO) severe pneumonia complicated by HIV and/or malnutrition, or severe hypoxemia.

STUDY HYPOTHESIS AND OBJECTIVES

• Study Hypotheses

The investigators hypothesize that bCPAP, compared to standard care, will reduce the mortality of Malawian children with WHO-defined severe pneumonia complicated by a severe co-morbidity (HIV-infection or HIV-exposure and/or severe malnutrition), or severe hypoxemia without a severe co-morbidity.

• Study Objectives

The broad objective of this study is to provide scientific evidence assessing the effectiveness of treatment with bCPAP for WHO severe childhood pneumonia for children 1-59 months of age in Malawi, Africa.

* Primary Objective 1

  • Determine the pneumonia mortality rate for bCPAP treatment, compared to standard of care, for children with WHO severe pneumonia.
* Primary Objective 2

  • Determine the pneumonia mortality rate for bCPAP treatment, compared to standard of care, for children with WHO severe hypoxemic pneumonia without co-morbidity (i.e., no HIV infection, no HIV-exposure, no severe malnutrition).
* Primary Objective 3

  • Determine the pneumonia mortality rate for bCPAP treatment, compared to standard of care, for children with WHO severe pneumonia and co-morbidity (i.e., HIV-infection or HIV-exposure and/or severe malnutrition).
* Secondary Objectives

  * Determine the pneumonia day 14 treatment failure rate for bCPAP treatment, compared to standard of care, for HIV-infected children with WHO severe pneumonia.
  * Determine the pneumonia day 14 treatment failure rate for bCPAP treatment, compared to standard of care, for HIV-exposed, uninfected children with WHO severe pneumonia.
  * Determine the pneumonia day 14 treatment failure rate for bCPAP treatment, compared to standard of care, for severely malnourished children with WHO severe pneumonia.
  * Determine the pneumonia day 14 treatment failure rate for bCPAP treatment, compared to standard of care, for severely hypoxemic children with WHO severe pneumonia.
  * Determine the proportion of children alive at day 30 phone follow up.
  * To investigate whether there may be differential treatment responses in certain baseline characteristics including but not limited to children with severe anemia, in those who test positive for malaria, in those with wheeze at baseline, in those with altered mental status, in those with digital auscultation-defined lung disease, and whether there is a differential treatment response by age.
  * To determine whether intervention arms have equivalent rates of adverse events as control arms.

ELIGIBILITY:
Inclusion Criteria:

* Meets World Health Organization (WHO) severe pneumonia criteria and is either Human Immunodeficiency Virus (HIV)-infected, HIV-exposed, severely malnourished, or has severe hypoxemia without HIV-infection, HIV-exposure, or severe malnutrition.

Exclusion Criteria:

* Any psychosocial condition or circumstance that, in the opinion of the investigators, would interfere with the conduct of the study. Prior participation in the study during a previous pneumonia diagnosis.

Ages: 1 Month to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 646 (Actual)
Dates: Start 2015-06-23 (Actual); Primary Completion 2018-04-28 (Actual); Study Completion 2018-04-28 (Actual)

PRIMARY OUTCOMES:
Pneumonia mortality | Participants followed for duration of hospital stay, an expected average of 7 days
  Proportion of in-hospital death in children with World Health Organization (WHO) severe pneumonia.

SECONDARY OUTCOMES:
Post-discharge mortality | 30 days after hospital discharge.
  Overall mortality 30 days after discharge.
Relapse | 30 days
  Proportion of children with a pneumonia cure but relapsed before day 30.
Treatment failure | 14 days
  Proportion of children failing treatment by day 14.

CONTACTS AND LOCATIONS:
Overall Officials: Eric D McCollum, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Salima District Hospital, Salima, Malawi

IPD SHARING:
Plan to Share IPD: Yes
Will be available upon request to principle investigator.

REFERENCES:
- [Derived] Sessions KL, Ruegsegger L, Mvalo T, Kondowe D, Tsidya M, Hosseinipour MC, Lufesi N, Eckerle M, Smith AG, McCollum ED. Focus group discussions on low-flow oxygen and bubble CPAP treatments among mothers of young children in Malawi: a CPAP IMPACT substudy. BMJ Open. 2020 May 12;10(5):e034545. doi: 10.1136/bmjopen-2019-034545. PMID 32404389
- [Derived] McCollum ED, Mvalo T, Eckerle M, Smith AG, Kondowe D, Makonokaya D, Vaidya D, Billioux V, Chalira A, Lufesi N, Mofolo I, Hosseinipour M. Bubble continuous positive airway pressure for children with high-risk conditions and severe pneumonia in Malawi: an open label, randomised, controlled trial. Lancet Respir Med. 2019 Nov;7(11):964-974. doi: 10.1016/S2213-2600(19)30243-7. Epub 2019 Sep 24. PMID 31562059
- [Derived] Sessions KL, Mvalo T, Kondowe D, Makonokaya D, Hosseinipour MC, Chalira A, Lufesi N, Eckerle M, Smith AG, McCollum ED. Bubble CPAP and oxygen for child pneumonia care in Malawi: a CPAP IMPACT time motion study. BMC Health Serv Res. 2019 Jul 31;19(1):533. doi: 10.1186/s12913-019-4364-y. PMID 31366394
- [Derived] Smith AG, Eckerle M, Mvalo T, Weir B, Martinson F, Chalira A, Lufesi N, Mofolo I, Hosseinipour M, McCollum ED. CPAP IMPACT: a protocol for a randomised trial of bubble continuous positive airway pressure versus standard care for high-risk children with severe pneumonia using adaptive design methods. BMJ Open Respir Res. 2017 Jun 30;4(1):e000195. doi: 10.1136/bmjresp-2017-000195. eCollection 2017. PMID 28883928